CLINICAL TRIAL: NCT01220908
Title: Evaluation of the PneumRx, Inc. Lung Volume Reduction Coil for the Treatment of Emphysema
Brief Title: Evaluation of the PneumRx Lung Volume Reduction Coil to Treat Emphysema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: PneumRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN0006
Record Dates: First submitted 2010-09-30; First posted 2010-10-14 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Emphysema
Keywords: LVRS (Lung Volume Reduction Surgery); LVRC (Lung Volume Reduction Coil); Emphysema; coil; RePneu
MeSH Terms: conditions — Emphysema | interventions — Pneumonectomy; Anterior Temporal Lobectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- permanent Coil(s) implant, QOL measure (Experimental): Coil implantation as treatment. Treatment is permanent implant.
  Interventions: Device: Lung Volume Reduction Coil (LVRC); Device: Coils

INTERVENTIONS:
Device: Lung Volume Reduction Coil (LVRC) — Implantation of Lung Volume Reduction Coil(s) (LVRC)
  Other Names: Lung Volume Reduction Surgery (LVRS); Lobectomy
Device: Coils — Lung Volume Reduction Coil(s)
  Other Names: Lung Volume Reduction Surgery (LVRS); Lobectomy

SUMMARY:
The objective of this study is to demonstrate the safety of the PneumRx Lung Volume Reduction Coil (LVRC) in a population of patients with emphysema. The PneumRx, Inc. LVRC is a used as a less invasive alternative to lung volume reduction surgery. The PneumRx LVRC is designed as an alternative to lung volume reduction surgery, potentially achieving the desired reduction in lung volume limiting the risks associated with major surgery, such as illness or death. This device is deployed through a bronchoscope and requires no incision.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 35 years of age
* unilateral or bilateral emphysema
* Patient has stopped smoking for a minimum of 8 weeks
* Read, understood and signed the Informed Consent form

Exclusion Criteria:

* Patient has a history of recurrent clinically significant respiratory infection
* Patient has an inability to walk >140 meters
* Patient has evidence of other disease that may compromise survival such as lung cancer, renal failure, etc
* Patient is pregnant or lactating
* Patient has clinically significant bronchiectasis
* Patient has had previous LVR surgery, lung transplant or lobectomy
* Patient has been involved in other pulmonary drug studies with 30 days prior to this study
* Patient has other disease that would interfere with completion of study, follow up assessments or that would adversely affect outcomes

Ages: 35 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-01; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Quality of Life Assessment. | Three + Months Follow-Up Visit
  Symptomatic improvement of Quality of Life as measured using the St. George's Respiratory Questionnaire (SGRQ)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk-Jan Slebos, MD, PhD, Principal Investigator — University Medical Center Groningen; Prof. Felix JF Herth, MD, PhD, Principal Investigator — Pneumology and Respiratory Care Medicine Thoraxklinik, University of Heidelberg
Locations (5):
- Germany (4):
  - Klinikum Donaustauf, Donaustauf
  - Asklepios, Gauting
  - Pneumology and Respiratory Care Medicine Thoraxklinik, University of Heidelberg, Heidelberg
  - Lungenklinik, Hemer
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Hartman JE, Klooster K, Gortzak K, ten Hacken NH, Slebos DJ. Long-term follow-up after bronchoscopic lung volume reduction treatment with coils in patients with severe emphysema. Respirology. 2015 Feb;20(2):319-26. doi: 10.1111/resp.12435. Epub 2014 Nov 23. PMID 25418910
- [Derived] Slebos DJ, Klooster K, Ernst A, Herth FJF, Kerstjens HAM. Bronchoscopic lung volume reduction coil treatment of patients with severe heterogeneous emphysema. Chest. 2012 Sep;142(3):574-582. doi: 10.1378/chest.11-0730. PMID 22116796